CLINICAL TRIAL: NCT02037152
Title: Smartphone-based Mindfulness Training for Chronic Pain: A Randomized Controlled Trial
Brief Title: Smartphone-based Mindfulness Training for Chronic Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with the software intervention, PI finished training and left UCSF.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBMT-CP-1; 13-10820 (Other: UCSF IRB)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Mobile applications; Mindfulness; Meditation; Telemedicine; Cellular phone; Pain Management; Therapy, computer-assisted
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist (No Intervention): Participants randomized to this arm are instructed that they will have access to the study intervention after four weeks. Waitlist group participants are prompted to answer weekly questionnaires.
- Active treatment (Experimental): The active treatment group will be instructed to use the app-guided "body scan" exercise daily for six days per week over a period of four weeks. The "body scan" includes 20 minutes of guided audio-- the pre-recorded voice of a narrator instructs the user to systematically direct attention to various parts of the body. Before and after each use of the body scan, users complete a single-item scale measuring pain intensity/distress. Users are prompted to complete all other questionnaires at weekly or four-week intervals. The app includes access to a graphical display showing changes in average pain level. Subjects also have access to a section of frequently asked questions about the practice.
  Interventions: Behavioral: Body scan exercise

INTERVENTIONS:
Behavioral: Body scan exercise — The "body scan" includes 20 minutes of guided audio-- the pre-recorded voice of a narrator instructs the user to systematically direct attention to various parts of the body. The audio content is adapted from the body scan exercises traditionally taught in evidence-based mindfulness interventions.
  Arms: Active treatment

SUMMARY:
The purpose of this study is to test a smartphone-based mindfulness training program for chronic pain. Research participants use a 20 minute app-guided audio program six days per week. The study hypothesis is that training in this technique over a period of four weeks will reduce pain interference with daily life activities. This study does not require any travel or in-person contact with research staff-- all elements of the study are completed on the participant's smartphone.

DETAILED DESCRIPTION:
This is a randomized, waitlist controlled trial. Smartphone users who download the research app complete an electronic informed consent before the app content is made available. Subjects meeting inclusion criteria are then prompted to complete baseline questionnaires. Submission of questionaires triggers randomization to one of two groups-- active treatment or waitlist. Subjects have equal chance of entering either group.

The active treatment group is instructed to use the app-guided "body scan" exercise daily for six days per week. The waitlist group is instructed that the research intervention will be made available to them in four weeks time. On a weekly basis, all subjects complete a Brief Pain Inventory scale. At the end of four weeks, subjects again complete a Brief Pain Inventory as well as the questionnaires measuring secondary outcomes. Upon completion of the control condition, waitlist subjects are invited to begin using the "body scan" exercise as described above. From this point forward, subjects receive the same protocol as the active treatment group. This study involves no face-to-face contact between participants and study investigators/staff.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Pain duration at least 3 months
* Access to smartphone

Exclusion Criteria:

* Pain from active cancer
* Pain from active cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Pain functional interference index | 4 weeks
  Change in pain functional interference index (part of Brief Pain Inventory questionnaire) during 4 week period

CONTACTS AND LOCATIONS:
Overall Officials: Ida Sim, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States